CLINICAL TRIAL: NCT01615081
Title: The Acute Effect of Malt Extract Versus Sucrose on the Response of Glucose and Insulin, Subjective Appetite Sensations and ad Libitum Energy Intake
Acronym: Harboe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, AAstrup, Professor, Dr Med, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B287
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Obesity; Diabetes
Keywords: Malt extract; carbohydrate; glucose response; insulin response; Appetite; Appetite regulating hormones
MeSH Terms: conditions — Obesity; Diabetes Mellitus | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sucrose solution (Active Comparator): 75 g sucrose (75 g carbohydrate) desolved in 750 ml water
  Interventions: Other: The acute effect of malt extract versus sucrose on the response of glucose and insulin, subjective appetite sensations and ad libitum energy intake
- Malt extract solution (Experimental): 183 g malt extract (corresponding to 75 g carbohydrate and 103 ml water) desolved in 647 ml water
  Interventions: Other: The acute effect of malt extract versus sucrose on the response of glucose and insulin, subjective appetite sensations and ad libitum energy intake

INTERVENTIONS:
Other: The acute effect of malt extract versus sucrose on the response of glucose and insulin, subjective appetite sensations and ad libitum energy intake — 2-arm crossover study for investigation of the effect of malt extract vs. sucrose on glucose, insulin, subjective appetite sensations and ad libitum energy intake.

SUMMARY:
Sucrose is the most used sweetener in beverage and foods in Denmark. Other sweeteners with other composition and amount of carbohydrates could be of interest in order to decrease the glucose and insulin responses after intake of a sweetened beverage/food. Malt extract has a sweet flavor but contains a different composition and amount of carbohydrates together with a small amount of protein compared to sucrose. Malt extract may therefore be a better alternative than sucrose as a sweetener due to a lower increase and more sustained blood glucose level. This could be of interest in relation to diabetes and appetite regulation but this is yet to be investigated.

Thus the objective is to investigate the effect of malt extract vs. sucrose on:

1. 3-hour change in the concentration of glucose and insulin
2. 3-hour change in subjective appetite sensations (Visual Analogue Scales, VAS scores)
3. Ad libitum energy intake

Design: 20 men will participate in the 2-way, randomized, double-blind crossover study. The test drinks is isocaloric with 75 g carbohydrates Test drinks: malt extract solution and sucrose solution (10%) Three-hour subjective appetite ratings and blood samples will be assessed every half-hour. Subsequently, the subjects will served an ad libitum lunch

ELIGIBILITY:
Inclusion Criteria:

* Healthy,
* BMI: 18.5-24.9 kg/m2,
* Weight stable (within +/- 3 kg) two months prior to study inclusion,
* Non-smoking,
* Nonathletic (< 10 h hard physical activity),

Exclusion Criteria:

* BMI > 25 kg/m2,
* Change in smoking status,
* Daily or frequent use of medication,
* Suffering from metabolic diseases,
* Suffering from psychiatric diseases,
* Suffering from any other clinical condition, which would make the subject unfit to participate in the study,
* Hemoglobin < 7.5 mmol/l.
* alcohol and drug abuse
* blood donation, 3mo prior to the present study and during study participation

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Acute 3-h changes from baseline in the postprandial concentration of glucose | Measured on 2 seperate test days in a crossover design. Each test day is seperated by >2 weeks. On each test day glucose is measured prior to the test drink (time 0) and 15, 30, 45, 60, 90, 120, 150, 180 minutes post intake
  Blood samples are taken prior to the test drink (baseline). After initiation of the test drink blood samples are collected at time 15, 30, 45, 60, 90, 120, 150, 180 minutes. Blood samples are analyzed for glucose.

SECONDARY OUTCOMES:
Acute 3-h changes from baseline in the postprandial concentration of insulin | Measured on 2 seperate test days in a crossover design. Each test day is seperated by >2 weeks. On each test day insulin is measured prior to the test drink (time 0) and 15, 30, 45, 60, 90, 120, 150, 180 minutes post intake
  Blood samples are taken prior to the test drink(baseline). After initiation of the test drink blood samples are collected at time 15, 30, 45, 60, 90, 120, 150, 180 minutes. Blood samples are analyzed for insulin.
Acute 3-h changes from baseline in subjective appetite sensations using visual analogue scales | Measured on 2 seperate test days in a crossover design. Each test day is seperated by >2 weeks. On each test day appetite sensations are measured prior to the test drink (time 0) and 15, 30, 45, 60, 90, 120, 150, 180 minutes post intake
  Assessment of subjective appetite sensations (visual analogue scales (VAS)) at time 0 (baseline - prior to the test meal) and at time 15, 30, 45, 60, 90, 120, 150, 180 minutes post intake.
  Measured subjective appetite sensations of hunger, satiety, prospective consumption, fullness, composite appetite score and sensory desires to something sweet, salty, rich in fat, or meat/fish.
Rating of the organoleptic quality of the test drinks | Measured on 2 seperate test days in a crossover design. Each test seperated by >2 weeks. On each test day after completion of the test drink (approximately) time 5 minutes post intake) subjects will rate the test drink
  After completion of the test drink the subjects will rate the organoleptic quality of the drink by visual analogue scales (VAS) in regard to appearance, smell, taste, after-taste, and general palatability.
Rating of the organoleptic quality of the ad libitum meal | Measured on 2 seperate test days in a crossover design. Each test seperated by >2 weeks. On each test day after completion of the ad libitum meal (approximately) time 15-20 minutes post intake) subjects will rate the ad libitum meal
  After completion of the adlibitum meal the subjects will rate the organoleptic quality of the meal by visual analogue scales (VAS) in regard to appearance, smell, taste, after-taste, and general palatability.
Subjective appetite sensations (visual analogue scales) after ad libitum meal | Measured on 2 seperate test days in a crossover design. Each test seperated by >2 weeks. After completion of the ad libitum meal subjects will rate their subjective sensation of appetite (approx 3.5-h post intake of test drink)
  After completion of the ad libitum meal the subjects will rate the subjective appetite sensations by visual analogue scales (VAS) in regard to sensation of hunger, satiety, prospective consumption, fullness, composite appetite score and sensory desires to eat something sweet, salty, rich in fat, or meat/fish.
change in body weight and composition (fat mass and fat free mass) | Measured on 2 seperate test days in a crossover design. Each test seperated by >2 weeks. On each test day body weight and composition is carried out prior to the test.
  body weight will be measured to the nearest 0.05 kg on a decimal scale. Body composition will be assessed by electric bioimpedance using an Animeter.
ad libitum energy intake (EI) | Measured on 2 seperate test days in a crossover design. Each test seperated by >2 weeks. EI was measured 180 min after intake of the test drink
  180 min after each test drink an ad libitum meal was served, and the total energy intake was recorded

CONTACTS AND LOCATIONS:
Overall Officials: Anne B Raben, Professor, Principal Investigator — Department of Human Nutrition, Faculty of Science, University of Copenhagen, Denmark
Locations (1):
- Department of Human Nutrition, Faculty of Science, University of Copenhagen, Frederiksberg, Denmark